CLINICAL TRIAL: NCT02982759
Title: Together We STRIDE (Strategizing Together Relevant Interventions for Diet and Exercise)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 8417; 1U01MD010540-01 (NIH); NCI-2018-02632 (Registry Identifier: NCI / CTRP); RG1001379 (Other: Fred Hutch / University of Washington Cancer Consortium)
Record Dates: First submitted 2016-11-30; First posted 2016-12-05 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comparison Arm (Other): The comparison group will receive 2 generic newsletters
  Interventions: Behavioral: Genetic Newsletters
- Intervention Arm (Experimental): The intervention arm will receive the multi-level intervention.
  Interventions: Behavioral: Multi-Level Intervention

INTERVENTIONS:
Behavioral: Multi-Level Intervention — The multi-level interventions will include activities at the individual level, family level, school level, and community level.
  Arms: Intervention Arm
Behavioral: Genetic Newsletters — The comparison will receive generic newsletters
  Arms: Comparison Arm

SUMMARY:
Obesity among Hispanic children in the Lower Yakima Valley of Washington State is alarmingly high. This study proposes to implement a comprehensive, multi-level intervention among children, families, the schools, and the community to combat this problem. The two year intervention will be measured by examining changes in children's body mass index.

DETAILED DESCRIPTION:
Childhood obesity rates in the Lower Yakima Valley of Washington State are alarming: 34% of youth are obese compared to the state average of 23%. A large proportion of those children are Hispanic; Hispanics represent 47% of the population in Yakima County and 67% of the population in the Lower Yakima Valley. In January 2013, the investigators study received a planning grant from the National Institute of Minority Health and Health Disparities to build and enhance community capacity and infrastructure on childhood obesity initiatives in the Lower Yakima Valley. This project began with the community as they expressed concern at the high incidence of obesity among Hispanic children in the Valley. In the ensuing two and a half years, the investigators and the community used community-based participatory research (CBPR) to 1) form a community advisory board (CAB); 2) build a Steering Committee; 3) conduct a comprehensive multi-level needs assessment; 4) develop and institute a pilot study; and 5) evaluate our activities. In response to RFA MD-15-010, the investigators and the community are now prepared to implement the intervention activities that were successful in our pilot study into a large-scale quasi-experimental intervention trial. The multi-level interventions will include activities at the individual level, family level, school level, and community level. Activities include distributing comic books to students about healthy eating and physical activity, a multi-generational level family intervention that teaches families about healthy eating and cooking skills as well as physical activity, a variety of school events to teach children about the food industry as well as encourage them to be physically activity at small intervals in the classroom, and community activities to foster the idea of the community being a healthy place for kids. The overall goal of this project is to continue to use a CBPR approach; in so doing, test the effectiveness of the comprehensive, multi-level intervention on reducing children's BMI z-scores, the primary endpoint. BMI z scores will be assessed by taking height and weight measures of the children at baseline, 12 months, and 24 months. This study will recruit and enroll a total of 900 Hispanic children in grades 3rd to 5th (ages 8-12 years) who attend the four elementary schools in the intervention community and the four elementary schools in the comparison community. Schools in both communities will be matched based on student standardized test scores, percent of students eligible to receive free or reduced-price lunch, and school size. Secondary outcomes include dietary patterns and accelerometer data of physical activity in a subgroup of 180 Hispanic children. Community participation in this project has been extraordinary and our letters of support indicate the communities' enthusiasm for this project.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic children in grade levels 3rd-5th (ages 8-12 years) who attend elementary schools in these two communities will be eligible to participate in the study.

Exclusion Criteria:

* Exclusion criteria include children with clinically-diagnosed dementia, terminal (<5 years) illness, major psychiatric illness, severe hearing impairment, and inability to move, which will be assessed during the distribution of the study recruitment packets to parents.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 888 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Body Mass Index z-score | 3 years

SECONDARY OUTCOMES:
Physical Activity with accelerometer | 3 years
Dietary Pattern with questionnaire | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Linda K Ko, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ko LK, Rillamas-Sun E, Kratz M, Jimenez E, Jang SH, Mendoza JA, Bishop S, Xiao L. A Multi-Level Intervention to Address Childhood Obesity in Rural Hispanic Communities. Obes Sci Pract. 2026 Jan 23;12(1):e70116. doi: 10.1002/osp4.70116. eCollection 2026 Feb. PMID 41584860
- [Derived] Ko LK, Rillamas-Sun E, Bishop S, Cisneros O, Holte S, Thompson B. Together We STRIDE: A quasi-experimental trial testing the effectiveness of a multi-level obesity intervention for Hispanic children in rural communities. Contemp Clin Trials. 2018 Apr;67:81-86. doi: 10.1016/j.cct.2018.02.013. Epub 2018 Mar 5. PMID 29501741